CLINICAL TRIAL: NCT03796195
Title: Does Stellate Ganglion Blockade (SGB) in Men Treated for Prostate Cancer Improve Hot Flashes? A Pilot Prospective Cohort Study
Brief Title: (SGB) in Men Treated for Prostate Cancer Improve Hot Flashes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment issues
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Walega, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00208657
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer; Hot Flashes
Keywords: Stelate Ganglion Block
MeSH Terms: conditions — Prostatic Neoplasms; Hot Flashes | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- .5% Bupivacaine (Experimental): Guided right sided stelate ganglion block using .5% bupivacaine (5mLs)
  Interventions: Drug: .5% Bupivacaine

INTERVENTIONS:
Drug: .5% Bupivacaine — Ultrasound guided right sided stelate ganglion block using .5% bupivacaine (5mLs)
  Other Names: Right sided stelate ganglion block (SGB)

SUMMARY:
Androgen Deprivation Therapy (ADT) is a critical component of advanced prostate cancer treatment but causes numerous adverse effects including decreased bone mass, decreased muscle mass, gynecomastia, erectile dysfunction, loss of sexual desire, depression, disordered sleep, urinary symptoms, and hot flashes (HF). HF are unpleasant paroxysmal episodes of flushing, sweating with vasodilation of the face, neck, and chest. These episodes can last for seconds to minutes and are often associated with night sweats, anxiety, and insomnia and have negative effects on quality of life.

Stellate ganglion blockade (SGB) with local anesthetic may be an effective treatment of HF in men on ADT, but has not been studied in any published clinical trials.

The stellate ganglion is a neural structure in the anterior cervical spine region and is part of the sympathetic nervous system. It has been injected safely in the practice of pain management for more than 50 years in cases of post herpetic neuralgia (shingles), complex regional pain syndrome (CRPS) and other painful neuropathies as well as some types of cardiac dysrhythmias.

Given the frequency and severity and interference of HF in men on ADT for prostate cancer, in addition to the negative effects HF impose on this patient population and a paucity of effective treatments, finding alternative treatments for HF in this population is needed.

ELIGIBILITY:
Inclusion Criteria:

1. Men with prostate cancer (with or without metastatic disease) on ADT for at least 2 months
2. Age less than 65 years
3. Body Mass Index (BMI) less than 32
4. Willingness to undergo image guided intervention
5. Greater than 28 hot flashes per week.

Exclusion Criteria:

1. Conditions that preclude SGB or sham intervention (e.g., anatomic abnormalities of the anterior neck or cervical spine; metastatic disease in or near the cervical spine; goiter;cardiac/pulmonary compromise; sleep apnea; acute illness/infection; coagulopathy or bleeding disorder; allergic reactions/contraindications to a local anesthetic or contrast dye)
2. Current treatment of prostate cancer with radium or chemotherapy
3. Use of treatments in the past two months that can affect HF (e.g., testosterone or androgen supplementation) Note: SSRIs, serotonin norepinephrine uptake inhibitors, and membrane stabilizers will be allowed but must be on stable unchanged dose for at least 8 weeks)
4. Inability to write, speak, or read in English

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with prostate cancer with bothersome hot flashes.
Enrollment: 1 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Walega, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez BD, Small BJ, Cases MG, Williams NL, Fishman MN, Jacobsen PB, Jim HSL. Sleep disturbance in men receiving androgen deprivation therapy for prostate cancer: The role of hot flashes and nocturia. Cancer. 2018 Feb 1;124(3):499-506. doi: 10.1002/cncr.31024. Epub 2017 Oct 26. PMID 29072790
- [Background] Dosani M, Morris WJ, Tyldesley S, Pickles T. The Relationship between Hot Flashes and Testosterone Recovery after 12 Months of Androgen Suppression for Men with Localised Prostate Cancer in the ASCENDE-RT Trial. Clin Oncol (R Coll Radiol). 2017 Oct;29(10):696-701. doi: 10.1016/j.clon.2017.06.009. Epub 2017 Jul 13. PMID 28712786
- [Background] Grunfeld EA, Hunter MS, Yousaf O. Men's experience of a guided self-help intervention for hot flushes associated with prostate cancer treatment. Psychol Health Med. 2017 Apr;22(4):425-433. doi: 10.1080/13548506.2016.1195504. Epub 2016 Jun 13. PMID 27294289
- [Background] Kouriefs C, Georgiou M, Ravi R. Hot flushes and prostate cancer: pathogenesis and treatment. BJU Int. 2002 Mar;89(4):379-83. doi: 10.1046/j.1464-4096.2001.01761.x. No abstract available. PMID 11872028
- [Background] Nishiyama T, Kanazawa S, Watanabe R, Terunuma M, Takahashi K. Influence of hot flashes on quality of life in patients with prostate cancer treated with androgen deprivation therapy. Int J Urol. 2004 Sep;11(9):735-41. doi: 10.1111/j.1442-2042.2004.00896.x. PMID 15379937
- [Background] Frisk J. Managing hot flushes in men after prostate cancer--a systematic review. Maturitas. 2010 Jan;65(1):15-22. doi: 10.1016/j.maturitas.2009.10.017. Epub 2009 Dec 4. PMID 19962840
- [Background] Trump DL. Commentary on "association of androgen deprivation therapy with cardiovascular death in patients with prostate cancer: a meta-analysis of randomized trials." Nguyen PL, Je Y, Schutz FA, Hoffman KE, Hu JC, Parekh A, Beckman JA, Choueiri TK, Department of Radiation Oncology, Dana-Farber Cancer Institute, Brigham and Women's Hospital, 75 Francis Street, Boston, MA 02115, USA: JAMA 2011;306(21):2359-66. Urol Oncol. 2012 Sep;30(5):746-7. doi: 10.1016/j.urolonc.2012.06.007. No abstract available. PMID 23021559
- [Background] Gavin AT, Donnelly D, Donnelly C, Drummond FJ, Morgan E, Gormley GJ, Sharp L. Effect of investigation intensity and treatment differences on prostate cancer survivor's physical symptoms, psychological well-being and health-related quality of life: a two country cross-sectional study. BMJ Open. 2016 Dec 19;6(12):e012952. doi: 10.1136/bmjopen-2016-012952. PMID 27993906
- [Background] Eziefula CU, Grunfeld EA, Hunter MS. 'You know I've joined your club... I'm the hot flush boy': a qualitative exploration of hot flushes and night sweats in men undergoing androgen deprivation therapy for prostate cancer. Psychooncology. 2013 Dec;22(12):2823-30. doi: 10.1002/pon.3355. Epub 2013 Jul 28. PMID 23893467

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | .5% Bupivacaine
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study closed early | 1

BASELINE CHARACTERISTICS:
Arm/Group | .5% Bupivacaine
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
Body Mass Index (kg/m^2) [Number; unit: (kg/m^2)] | 25
Baseline Hot Flash-Related Daily Interference Scale (HFRDIS) [Number; unit: score on a scale] — HFRIDS is a 10 question survey scored on a scale of 0=no interference and 10=high interference.
  Questions inquire about work, social activities, leisure activities,sleep, mood,concentratoin, relationship with others, sexuality,enjoyment of life and overqll quality of life. Low score=0 is the lowest interference score and the highest interference score is 100.
  score on a scale | 48
Baseline mean daily hot flashes [Number; unit: Hot flashes/day] — Baseline mean daily hot flashes reported by subject using daily diary.
  Hot flashes/day | 9.78
PROMIS SF4a Sleep Score [Number; unit: Score on a scale] — PROMIS SF4a (sleep) Patient Reported Outcomes Measurement Information System. The PROMIS SF4a is a 4 item questionnaire that queries sleep duration, quality and interruption. This instrument accesses self reported perceptions of sleep quality. sleep depth and restoratoin associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of satisfaction with sleep. The 4 items are scored 1-5 where 1 is good quality and 5 is poor quality for a total score range of 4 (good quality) to 20 (poor quality).
  Score on a scale | 11

OUTCOME MEASURES:

1. Primary Outcome: Hot Flash Frequency Change Baseline to 3 Months After Treatment.
Description: Change in mean daily hot flashes using a self-report hot flash diary from baseline to 3 months after stellate ganglion block.
Time Frame: 3 months after SGB procedure
Measure: Number; unit: Hot flashes/day
Arm/Group | .5% Bupivacaine
Number analyzed (Participants) | 1
Hot flashes/day | -1.78

2. Secondary Outcome: Change in Hot Flash Severity Baseline to 3 Months After Stellate Ganglion Block
Description: The change in hot flash severity (hot flash frequency x hot flash intensity) between baseline and 3 months after SGB. Hot flash severity is determined using the mean frequency= ((Fmo+Fse))7 where FMi, Fmo and Fse are the weekly total number of mild, moderate or severe HF events. The mean severity= (Fmi+2x Fmo + 3 x Fse)/7 where FMI, Fmo and Fse are the weekly total number of mild, moderate or severe/very severe hot flash events in the case of mean severity, frequency of mild vasomotor symptoms is not counted at baseline.
Time Frame: 3 months after stellate ganglion block
Measure: Number; unit: Score on a scale
Arm/Group | .5% Bupivacaine
Number analyzed (Participants) | 1
Score on a scale | -55.94

3. Secondary Outcome: PROMIS SF4a Score 4 Weeks After Stellate Ganglion Block.
Description: PROMIS SF4a (sleep) Patient Reportee Outcomes Measurement Information System. The PROMIS SF4a is a 4 item questionnaire that queries sleep duration, quality and interruption. This instrument accesses self reported perceptions of sleep quality, sleep depth and restoratoin associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy and satisfaction with sleep. The 4 items are scored 1-5 where 1 is good quality and 5 is poor quality for a total score range of 4 (good quality) to 20 (poor quality).
Time Frame: 4 weeks after stellate ganglion block
Measure: Number; unit: Score on a scale
Arm/Group | .5% Bupivacaine
Number analyzed (Participants) | 1
Score on a scale | 8

4. Secondary Outcome: Patient Global Impression of Change Score (PGIC)
Description: The PGIC assesses the participants improvement in hot flashes from the time of the stellate ganglion block to 4 weeks after the procedure. The PGIC queries how much the hot flashes have improved on a scale of 1 (very much improved) to 7 (very much worse).
Time Frame: 4 weeks after stellate ganglion block
Measure: Number; unit: Score on a scale
Arm/Group | .5% Bupivacaine
Number analyzed (Participants) | 1
Score on a scale | 4

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for 4 weeks after stellate ganglion block procedure.
Description: Data obtained by telephone call up to 4 weeks post stellate ganglion block procedure.
Arm/Group | .5% Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study was closed early for slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT03796195/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT03796195/ICF_001.pdf